CLINICAL TRIAL: NCT06413394
Title: The Effect of Virtual Reality Supported Environmental Ethics Approaches Education on Nurse's Empathy and Environmental Ethics Awareness Levels
Brief Title: Virtual Reality, Empathy and Environmental Ethics.
Status: Completed | Type: Observational
Sponsor: Ardahan University (Other)
Responsible Party: Sponsor
Other Study IDs: ArdahanUniversiserhatduzenci01
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Virtual Reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Virtual reality supported environmental education group: virtual reality supported environmental education group
  Interventions: Other: environmental education
- The group that will not receive virtual reality-supported environmental education: the group that will not receive virtual reality-supported environmental education
  Interventions: Other: environmental education
- Control group: control group

INTERVENTIONS:
Other: environmental education — environmental education
  Groups: The group that will not receive virtual reality-supported environmental education; Virtual reality supported environmental education group

SUMMARY:
Environmental ethics is a sub-branch of ethics that determines moral values and principles towards the environment. It is the common responsibility of all humanity to improve and protect the environment/nature and to hand it over to the next generations. For this reason, every segment of society should have environmental ethics awareness. Empathy is an important concept in raising awareness of environmental ethics. It is stated that the awareness of environmental ethics is also developed in people who have developed empathy skills. For this reason, it is recommended to create training programs that enable people to develop their empathy skills. The formation and establishment of environmental ethics awareness in people can prevent the occurrence of environmental problems. This can be achieved by providing an effective environmental education. Technological developments such as virtual reality can be used in environmental education. Virtual reality technologies are called empathy machines as they create a sense of presence in users. For this reason, the perception of presence in virtual reality and being included in the narrative are effective in developing empathy in the person. It is stated that the perspectives acquired in virtual reality develop empathy and encourage behaviors in favor of society in a few weeks. Virtual reality technologies are useful for us researchers, both in terms of developing empathy towards environmental problems and creating awareness of environmental ethics as an educational tool. For this reason, in this study, the effect of virtual reality supported environmental education on nurses' empathy and environmental ethics awareness levels was tried to be examined with a quasi-experimental research.

DETAILED DESCRIPTION:
RESEARCH DESIGN This research is a three-arm randomized controlled experimental study conducted prospectively to compare the effect of virtual reality-supported environmental education on nurses' environmental ethics approaches and empathy levels.

LOCATION AND CHARACTERISTICS OF THE STUDY This research was conducted at a State Hospital located in a province in the Eastern Anatolia Region between 01.10.2022 and 31.04.2023. The hospital consists of primary adult intensive care, secondary adult intensive care, secondary neonatal intensive care, six-bedded wards, operating theatre service, emergency department, palliative care unit, dialysis unit, and outpatient care service. The working hours of the hospital are organized in two shifts, 08.00-16.00 and 16.00-08.00, or 24 hours (full day).

POPULATION AND SAMPLE SELECTION The research was conducted with 91 nurses who volunteered to participate from among 101 nurses working at a State Hospital in a province in the Eastern Anatolia Region between 01.10.2022 and 31.04.2023. The total sample size was calculated as 90 (n=90) using G-POWER program with .4 (Cohen) effect size, 92% power, and .05 error margin based on percentage measurement values of the methods to be studied obtained from literature review (Faul et al., 2007). Considering possible losses, 33 nurses were planned to be included in each group, and randomization was performed over 91 nurses. None of the nurses included in the study met the exclusion criteria, and the study was concluded with 91 nurses.

Inclusion Criteria for the Sample

* Being a nurse working at the relevant State Hospital
* Volunteering to participate in the research
* Not having received virtual reality-supported environmental education before

Exclusion Criteria for the Sample

* Not being a nurse working at the relevant State Hospital
* Not volunteering to participate in the research
* Having received virtual reality-supported environmental education before

Criteria for Withdrawal from the Sample

* Being absent at any time during the research process
* Not completing the environmental education

Dependent and Independent Variables of the Study The main independent variable of the study is virtual reality-supported environmental education. Other sub-variables are data obtained through the "Nurse Introduction Form" and the "Empathy Level Determination Scale." The dependent variable of the study is data obtained through the "Environmental Ethics Approaches Scale."

FORMS AND SCALES USED IN DATA EVALUATION The "Nurse Introduction Form," "Empathy Level Determination Scale," and "Environmental Ethics Approaches Scale" were used in the study

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in ardahan state hospital

Exclusion Criteria:

* Nurses not working in ardahan state hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Scale for Environmental Ethics Approaches | 15/11/2022-31/12/2022
  Scale for environmental ethics approaches pre-test
Scale for Environmental Ethics Approaches | 16/02/2023-28/03/2023
  Scale for environmental ethics approaches post-test
Adaptation of Empathy Quotient (EQ) Scale | 15/11/2022-31/12/2022
  Adaptation of Empathy Quotient (EQ) Scale pre-test
Adaptation of Empathy Quotient (EQ) Scale | 16/02/2023-28/03/2023
  Adaptation of Empathy Quotient (EQ) Scale post-test

CONTACTS AND LOCATIONS:
Overall Officials: Bahanur Malak Akgün, Principal Investigator — Ardahan University
Locations (1):
- Ardahan Devlet Hastanesi, Ardahan, Centrium, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
gender, total working time, age, marital status